CLINICAL TRIAL: NCT07168798
Title: Evaluation of SpO2 Accuracy in Children With Various Skin Color
Brief Title: SpO2 Accuracy in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Nihon Kohden (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 25-023147
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypoxemia
Keywords: Spo2; Pulse oximetry; skin tone
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled subjects: Subjects who meet the enrollment criteria
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — OLV-4201 pulse oximeter with sensors: TL-272T3, TL-274T3 and TL-273T3

SUMMARY:
Evaluation of SpO2 Accuracy in Children with Various Skin Color

DETAILED DESCRIPTION:
Pulse oximeters, which estimate blood oxygen levels, are routinely utilized for monitoring. However, research has shown that these devices may provide higher readings for individuals with darker skin tones as compared to individuals with lighter skin tones. This inaccuracy can result in unnoticed or untreated low oxygen levels, particularly affecting racial and ethnic minorities. It is beneficial for patients and healthcare providers to evaluate the accuracy of pulse oximeter oxygen saturation (SpO2) readings from pulse oximeters sold in the U.S. This study test the Nihon Kohden pulse oximeter and SpO2 sensors in neonatal and pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 - 12 who are admitted to the CICU with or plan to have an indwelling arterial line for standard care

Exclusion Criteria:

* Patients with elevated levels of methemoglobin and carboxyhemoglobin, or anemia.
* Patients with prolonged hypotension at the time of enrollment.
* Patients with ductal-dependent congenital cardiac disease.

Ages: 0 Days to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
SpO2 accuracy | 24 hours
  Evaluate the accuracy of Nihon Kohden SpO2 in measuring blood oxygen levels in children with varying skin tones

SECONDARY OUTCOMES:
SpO2 to SaO2 agreement | 24 hours
  Evaluate the agreement between Nihon Kohden SpO2 and arterial oxygen saturation (SaO2) in children with varying skin tones

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Y Naim, M.D., MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Proprietary information

REFERENCES:
- [Result] Sjoding MW, Dickson RP, Iwashyna TJ, Gay SE, Valley TS. Racial Bias in Pulse Oximetry Measurement. N Engl J Med. 2020 Dec 17;383(25):2477-2478. doi: 10.1056/NEJMc2029240. No abstract available. PMID 33326721